CLINICAL TRIAL: NCT06593158
Title: Effect of Parent-delivered Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) in Young Children With Cerebral Palsy in Vietnam
Brief Title: Parent-delivered HABIT-ILE in Young Children With Cerebral Palsy in Vietnam
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Parent-delivered HABIT-ILE
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy
Keywords: HABIT-ILE; Cerebral Palsy; Caregiver -delivered; Intensive therapy; Home rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The trial will be a single-blind, randomized controlled trial. Participants will be randomly assigned to one of two groups: HABIT-ILE Camp with Caregivers or HABIT-ILE at Home with Caregivers. Both groups will have longitudinal assessments two weeks before baseline, at baseline, at the end of the two-weeks intervention, and 3 months after baseline.
Who Masked: Outcomes Assessor
Masking Description: The primary outcomes: The Gross Motor Function Measure (GMFM-66), Melbourne Assessment 2 will be videotaped, and the scoring will be done by blind trained examinors.
  In secondary outcomes: ACTIVLIM-CP-WA, PEDI, COPM, WHOQOL-Bref will be answered by the caregivers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE at Camp with Caregivers (Active Comparator)
  Interventions: Behavioral: Parent-delivered Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) for CP children at camp with the guidance and supervision of experts.
- HABIT-ILE at Home with Caregivers (Active Comparator)
  Interventions: Behavioral: Parent-delivered Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) for CP children at home with the online guidance and supervision of experts.

INTERVENTIONS:
Behavioral: Parent-delivered Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) for CP children at camp with the guidance and supervision of experts. — * The caregivers delivering HABIT-ILE therapy at camp will follow the same principles as the usual HABIT-ILE. The therapy will take place in a rehabilitation center, and caregivers will provide therapy during the sessions, coached by trained supervisors on site
  * The intervention day will then take place, lasting for 5 hours with the constant presence of supervisors. This will be divided into two sessions: a 3-hour intervention in the morning followed by a lunch break, and a 2-hour intervention in the afternoon.
  Arms: HABIT-ILE at Camp with Caregivers
Behavioral: Parent-delivered Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) for CP children at home with the online guidance and supervision of experts. — * The caregivers delivering HABIT-ILE therapy at home will follow the same principles as the usual HABIT-ILE. The therapy will take place at children's home, caregivers will provide therapy during the sessions, coached by trained supervisors online
  * The intervention day will then take place, lasting for 5 hours with the supervisors through online setting. This will be divided into two sessions: a 3-hour intervention in the morning followed by a lunch break, and a 2-hour intervention in the afternoon.
  Arms: HABIT-ILE at Home with Caregivers

SUMMARY:
This study will use a randomized controlled trial design with a longitudinal baseline to assess the effectiveness of Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) on motor function and the ability to perform daily activities in Vietnamese children with cerebral palsy, specifically through a caregiver-delivered approach. Participants will be randomly assigned to one of two groups: HABIT-ILE at Camp with Caregivers and HABIT-ILE at Home with Caregivers. The study aims to determine whether a caregiver-delivered intervention will be effective compared to the "no intensive" phase and whether on-site intervention with the constant presence of supervisors may have additional effects.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of non-progressive early onset neuromotor disorders that affect the developing brain of the fetus or infant. Motor disorders in CP are often accompanied by sensory, perceptual, cognitive, communicative, and behavioural disorders, and secondary musculoskeletal problems. CP is characterized by impairment in gross motor function involving large muscles which perform daily activities such as walking, standing, running, jumping and fine motor function involving small muscles in the hand and wrist which perform flexible hand and finger grip activities, communication ability. The purpose of rehabilitation in children with CP is to minimize the impact of physical disability, to improve independence in the community and to improve the quality of life of children and their families.

Traditionally, CP was managed through neurorehabilitation based on neurodevelopmental methods. However, the effectiveness of these methods is still being hotly debated. In contrast, there is evidence that intensive therapy based on motor skill learning is more effective in creating functional and neuroplastic changes. Intensive therapy is a high-intensity program completed daily for several weeks, focusing on repetitive tasks with gradually increasing difficulty towards functional goals identified by the child and the child's caregiver. Hand-arm bimanual intensive therapy including lower extremities (HABIT-ILE) has shown improvement in motor and functional outcomes in children with CP. HABIT-ILE therapy is recommended in high-income countries (HIC) in the form of camps where children practice continuously for a short period (2 weeks), totalling 50-90 hours in a treatment session with therapists. In Vietnam, rehabilitation is not widely accessible, possibly due to high treatment costs and a lack of treatment facilities and staff. Recognizing the potential of HABIT-ILE therapy and the practical context of Vietnam, in this study, we aim to apply Parent-delivered HABIT-ILE and explore the effectiveness of this therapy on children with CP in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Cerebral palsy
* Type of Cerebral palsy: Bilateral cerebral palsy
* Level of gross motor function: level II to IV of GMFCS E& R
* Level of manual ability: level I to IV of mini- MACS
* Environmental factors: Having caregiver support during the study (availability of a caregiver for 5h per day during two weeks of therapy)
* Age of children: 2 to 6 years old

Exclusion Criteria:

* The child has uncontrolled seizures.
* The child has visual impairment that could interfere with the assessment and treatment.
* The child has severe cognitive problems, unable to understand or be interested in simple games
* Other intensive therapy or surgery/medical intervention that could interfere with study results in the past 6 months and during the study period (e.g. botulinum toxin, etc).

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure -66 (GMFM- 66) | Two weeks before baseline, at baseline, at the end of the two-weeks intervention, and 3 months after baseline
  The GMFM-66 is a 66-item scale that is divided into five aspects of gross motor function: lying and rolling, sitting, crawling, and kneeling, standing, and walking, running, and jumping. All items are arranged in order of difficulty and have a common unit of change from 0 to 100
Melbourne Assessment 2 | Two weeks before baseline, at baseline, at the end of the two-weeks intervention, and 3 months after baseline
  - The Melbourne Assessment 2 (MA2) is a reliable and valid tool used to assess upper limb movement quality in children aged 2.5 to 15 with neurological impairments. It evaluates four key areas: range of motion, accuracy of reaching and placement, dexterity of grasp, release, and manipulation, and fluency of movement. The 14-item test involves children reaching for, grasping, releasing, and manipulating simple objects while their performance is video recorded for later scoring.

SECONDARY OUTCOMES:
ACTIVLIM-CP-WA questionnaire | Two weeks before baseline, at baseline, at the end of the two-weeks intervention, and 3 months after baseline
  ACTIVLIM-CP-WA questionnaire measures global performance of daily life activities in children with cerebral palsy (CP). The ACTIVLIM-CP-WA was built on the parents' perception and involves 31 items covering the domain of self-care, mobility and domestic life of the International Classification of Functioning, Disability and Health, Child, and Youth version (ICF-CY). The 31 items of the ACTIVLIM-CP-WA include 21 items for preschoolers (2 to 6 years), 23 items for children aging 6 to 12 years and 19 items for teens (12 to 19 years). Parents are instructed to estimate their child's difficulty in performing the activities related to the age of the child, as mentioned in the questionnaire, on three-level responses: Impossible (the child is unable to perform the activity alone), Difficult (the child is able to perform the activity alone, but experiences some difficulties), Easy (the child is able to perform the activity alone, without any difficulty).
Paediatric Evaluation of Disability Inventory (PEDI) | Two weeks before baseline, at baseline, at the end of the two-weeks intervention, and 3 months after baseline
  PEDI is an interview-based tool that assesses functional performance in children. It is divided into three parts. In part I, this tool assesses in Functional kills of children with some domains such as: Self Care, Mobility, Social Function. Each domain evaluates specific tasks including feeding, dressing, walking, and communicating with others. It is scored on a four-point scale: 0 - unable, 1 - capable. In part II and III, this tool assesses in Caregiver Assistance with some domain such as: Self-Care, Mobility, Social Function. Using a 5-point scale: 5 - independence, 4 - supervision, 3 - average assistance, 2 - minimal assistance, 1 - maximum assistance, 0 - complete assistance.
The Canadian Occupational Performance Measure (COPM) | Two weeks before baseline, at baseline, at the end of the two-weeks intervention, and 3 months after baseline
  COPM is a client-centred outcome measure that allows individuals to identify and prioritize daily issues that limit their participation in everyday life. The measure focuses on the performance of activities in all areas of life, including self-care, leisure, and productivity to identify and prioritize daily issues that limit their participation in everyday life. 5 of the most important goals are then further assessed using a 10-point scale for performance and satisfaction.
WHOQOL-BREF | Two weeks before baseline, at baseline, at the end of the two-weeks intervention, and 3 months after baseline
  WHOQOL-BREF is a self-administered questionnaire that includes 26 questions about individuals' perceptions of their health and mental state in the two weeks prior. Answers to the questions are scored on a 1-5 Likert scale, where 1 represents "disagree" or "strongly disagree" and 5 represents "strongly agree" or "extremely agree". WHOQOL-BREF consists of four domains, each with specific aspects: physical health, psychological, social relationships, environment.

IPD SHARING:
Plan to Share IPD: No